CLINICAL TRIAL: NCT00423696
Title: Phase II Randomized Study of First-Line Therapy Comprising Bevacizumab and Irinotecan Hydrochloride, Leucovorin Calcium, and Fluorouracil (FOLFIRI) Versus Bevacizumab and Irinotecan Hydrochloride and Capecitabine (XELIRI) in Patients With Unresectable Metastatic Colorectal Cancer [ACCORD]
Brief Title: Bevacizumab and Combination Chemotherapy as First-Line Therapy in Treating Patients With Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000523435; FRE-FNCLCC-ACCORD-13-0503 (Other: UNICANCER); EU-20666 (Registry Identifier: European Union); 2005-000070-43 (EudraCT Number)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bevacizumab + FOLFIRI (Experimental)
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium
- bevacizumab + XELIRI (Experimental)
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: irinotecan hydrochloride

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine
  Arms: bevacizumab + XELIRI
Drug: fluorouracil
  Arms: bevacizumab + FOLFIRI
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
  Arms: bevacizumab + FOLFIRI

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with combination chemotherapy may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective when given together with bevacizumab in treating patients with colorectal cancer.

PURPOSE: This randomized phase II trial is studying bevacizumab to compare how well it works when given together with two different combination chemotherapy regimens as first-line therapy in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival at 6 months in patients with unresectable metastatic colorectal cancer treated with first-line therapy comprising bevacizumab and irinotecan hydrochloride, leucovorin calcium, and fluorouracil (FOLFIRI) vs bevacizumab and irinotecan hydrochloride and capecitabine (XELIRI).

Secondary

* Compare the toxicities of these regimens in these patients.
* Compare the objective response rate and duration of response in patients treated with these regimens.
* Compare the tumor control in patients treated with these regimens.
* Compare the progression-free and overall survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to participating center, WHO performance status (0 or 1 vs 2), age (< 65 years vs ≥ 65 years), and number of metastatic sites (1 vs ≥ 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients may then continue to receive bevacizumab alone every 2 weeks in the absence of disease progression.
* Arm II: Patients receive bevacizumab IV over 30-90 minutes and irinotecan hydrochloride IV over 90 minutes on day 1 and oral capecitabine on days 1-14. Treatment repeats every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity. Patients may then continue to receive bevacizumab alone every 3 weeks in the absence of disease progression.

Quality of life is assessed periodically.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 144 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Unresectable metastatic disease
* Measurable disease
* No CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9 g/dL (transfusion allowed)
* INR < 1.5
* Alkaline phosphatase < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* AST and ALT < 2.5 times ULN (5 times ULN if liver metastases are present)
* Creatinine clearance > 30 mL/min
* Urine protein < 2+ OR ≤ 1 g/L by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindications to study therapy
* No gastrointestinal or duodenal ulcers
* No AIDS
* No serious illness, active infection, or other serious condition that would preclude study therapy
* No coagulation problem
* No bleeding diathesis
* No sensitivity to Chinese hamster ovarian cells or other recombinant human antibodies
* No severe renal insufficiency
* No uncontrolled hypertension
* No active or severe cardiovascular conditions, including the following:

  * Cerebrovascular accident
  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV cardiac insufficiency
  * Severe cardiac arrhythmia (even if treated)
* No primitive stenosis or symptomatic peritoneal carcinosis causing a risk of intestinal subocclusion or occlusion
* No nonhealing wound or fracture
* No prior thromboembolic disease
* No other cancer within the past 2 years except for basal cell skin cancer or carcinoma in situ of the uterine cervix
* No geographical, social, or psychological condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease
* At least 6 months since prior adjuvant chemotherapy (fluorouracil with or without oxaliplatin)

  * No prior adjuvant chemotherapy comprising irinotecan hydrochloride with or without bevacizumab
* At least 28 days since prior major surgery
* Prior radiotherapy allowed except to target lesions
* At least 10 days since prior anticoagulants
* No concurrent chronic acetylsalicylic acid (at doses > 325 mg/day)
* No other concurrent investigational therapy
* No other concurrent anticancer therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-03-23 (Actual); Primary Completion 2008-07-28 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months

SECONDARY OUTCOMES:
Percentage of objective responses
Percentage of stable disease responses
Duration of objective response and stable disease
Progression-free survival
Overall survival
Toxicities
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ducreux, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (15):
- France (15):
  - C.H.U. de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Polyclinique des Quatre Pavillons, Lormont
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Hopital, Paris
  - Polyclinique Francheville, Périgueux
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Malka D, Boige V, Jacques N, Vimond N, Adenis A, Boucher E, Pierga JY, Conroy T, Chauffert B, Francois E, Guichard P, Galais MP, Cvitkovic F, Ducreux M, Farace F. Clinical value of circulating endothelial cell levels in metastatic colorectal cancer patients treated with first-line chemotherapy and bevacizumab. Ann Oncol. 2012 Apr;23(4):919-27. doi: 10.1093/annonc/mdr365. Epub 2011 Aug 8. PMID 21825101
- [Derived] Antoun S, Bayar MA, Dyevre V, Lanoy E, Smolenschi C, Ducreux M. No evidence for changes in skeletal muscle mass or weight during first-line chemotherapy for metastatic colorectal cancer. BMC Cancer. 2019 Aug 28;19(1):847. doi: 10.1186/s12885-019-6086-2. PMID 31462288